CLINICAL TRIAL: NCT02247401
Title: An Open-Label Study to Evaluate the Safety and Efficacy of the Coadministration of ABT-450/Ritonavir/ABT-267 (ABT-450/r/ABT-267) With Ribavirin (RBV) in Adults With Chronic Hepatitis C Virus Genotype 4 Infection in Egypt
Brief Title: Coadministration of ABT-450/Ritonavir/ABT-267 (ABT-450/r/ABT-267) With Ribavirin (RBV) in Adults With Genotype 4 (GT4) Hepatitis C Virus (HCV) in Egypt
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M14-250
Record Dates: First submitted 2014-09-19; First posted 2014-09-25 (Estimated); Results first posted 2017-07-27 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: HCV; Hepatitis C Infection; Genotype 4
Keywords: Genotype 4; non-responder; treatment experienced; HCV; naive; relapser; hepatitis infection; compensated cirrhosis; hepatitis c; Cirrhosis; Egypt; null responder; partial responder
MeSH Terms: conditions — Hepatitis C; Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm A (Active Comparator): ABT-450/r/ABT-267 (paritaprevir/ritonavir/ombitasvir; 2 direct acting antiviral agent [DAA]) plus Ribavirin (RBV) for 12 weeks in treatment-naïve and treatment-experienced (with pegylated interferon and ribavirin) participants without cirrhosis.
  Interventions: Drug: 2 DAA; Drug: RBV
- Arm B (Active Comparator): ABT-450/r/ABT-267 plus RBV for 12 weeks in treatment-naïve and treatment-experienced (with pegylated interferon and ribavirin) participants with compensated cirrhosis.
  Interventions: Drug: 2 DAA; Drug: RBV
- Arm C (Active Comparator): ABT-450/r/ABT-267 plus RBV for 24 weeks in treatment-naïve and treatment-experienced (with pegylated interferon and ribavirin) participants with compensated cirrhosis.
  Interventions: Drug: 2 DAA; Drug: RBV

INTERVENTIONS:
Drug: 2 DAA — ABT-450/r/ABT-267 tablets
Drug: RBV — Ribavirin tablets

SUMMARY:
This study evaluates the efficacy and safety of ABT-450/r/ABT-267 with RBV in treatment-naive and treatment-experienced HCV GT4 subjects without or with compensated cirrhosis.

DETAILED DESCRIPTION:
Non-cirrhotic subjects were directly enrolled into Arm A. Cirrhotic subjects were randomized to either Arm B (12 weeks of treatment) or Arm C (24 weeks of treatment).

ELIGIBILITY:
Inclusion Criteria:

* Chronic hepatitis C, genotype 4-infection (hepatitis C virus [HCV] ribonucleic acid [RNA] level greater than 1,000 IU/mL at Screening)
* Subjects must meet one of the following:

  * Treatment-naive: Subject has never received antiviral treatment for HCV infection OR
  * Treatment Experienced (Prior null responders, Partial responders or Relapsers to pegylated-interferon [pegIFN]/RBV);
* Females must be post-menopausal, of non-child bearing potential or practicing specific forms of birth control
* In substudy 1, demonstrated absence of liver cirrhosis as confirmed by liver biopsy or Fibroscan
* In substudy 2, evidence of liver cirrhosis as confirmed by liver biopsy or Fibroscan with Child-Pugh score less than or equal to 6 at Screening and confirmed absence of hepatocellular carcinoma

Exclusion Criteria:

* Females who are pregnant or breastfeeding
* Positive screen for hepatitis B Surface antigen or anti-Human Immunodeficiency virus antibody
* HCV genotype performed during screening indicating unable to genotype or co-infection with any other HCV genotype
* abnormal laboratory tests
* self-reports current drinking more than 2 drinks per day
* current enrollment in another investigational study
* previous treatment with a direct acting antiviral agent (DAA) containing regimen
* In substudy 1, evidence of liver cirrhosis
* In substudy 2, evidence of current or past Child-Pugh B or C classification and confirmed presence of hepatocellular carcinoma

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2014-11-04; Primary Completion 2016-08-01 (Actual); Study Completion 2016-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Kopecky-Bromberg, PhD, Study Director — AbbVie

REFERENCES:
- [Background] Waked I, Shiha G, Qaqish RB, Esmat G, Yosry A, Hassany M, Soliman R, Mohey MA, Allam N, Zayed N, Asselah T, Hall C, Redman R, Mobashery N, Doss W. Ombitasvir, paritaprevir, and ritonavir plus ribavirin for chronic hepatitis C virus genotype 4 infection in Egyptian patients with or without compensated cirrhosis (AGATE-II): a multicentre, phase 3, partly randomised open-label trial. Lancet Gastroenterol Hepatol. 2016 Sep;1(1):36-44. doi: 10.1016/S2468-1253(16)30002-4. Epub 2016 Jun 16. PMID 28404110

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Safety population: All participants who received at least one dose of study drug.
Groups:
- Arm A: ABT-450/r/ABT-267 (paritaprevir/ritonavir/ombitasvir; 2 DAA) plus Ribavirin (RBV) for 12 weeks in treatment-naïve and treatment-experienced (with pegylated interferon and ribavirin) participants without cirrhosis.
Period: Overall Study
Arm/Group | Arm A | Arm B | Arm C
Started | 100 | 31 | 29
Completed | 94 | 29 | 27
Not Completed | 6 | 2 | 2
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 1 | 1
Not completed — Lost to Follow-up | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Arm C | Total
Number analyzed (Participants) | 100 | 31 | 29 | 160
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.6 (13.14) | 57.3 (6.48) | 55.8 (8.02) | 51.6 (11.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 2 | 7 | 39
  Male | 70 | 29 | 22 | 121

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response 12 Weeks Post-treatment (SVR12) in Each Treatment Arm
Description: SVR12 was defined as hepatitis C virus ribonucleic acid (HCV RNA) level less than the lower limit of quantification (< LLOQ) 12 weeks after the last dose of study drug.
Time Frame: 12 weeks after last dose
Population: Intent-to-treat population: all participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A | Arm B | Arm C
Number analyzed (Participants) | 100 | 31 | 29
percentage of participants | 94.0 [87.5 to 97.2] | 96.8 [83.8 to 99.4] | 93.1 [78.0 to 98.1]

2. Primary Outcome: Number of Participants With Adverse Events
Description: An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. The investigator assessed the relationship of each event to the use of study drug as either reasonable possibility or no reasonable possibility. A serious adverse event (SAE) is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment, may jeopardize the subject and may require medical or surgical intervention to prevent any of the outcomes listed above. Treatment-emergent events (TEAEs/TESAEs) are defined as any event that began or worsened in severity after the first dose of study drug. For more details on adverse events please see the Adverse Event section.
Time Frame: Screening until 30 days after last dose
Population: Safety Population: all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B | Arm C
Number analyzed (Participants) | 100 | 31 | 29
Participants | 80 | 26 | 25

3. Secondary Outcome: Percentage of Participants With On-treatment Virologic Failure in Each Treatment Arm
Description: On-treatment virologic failure was defined as quantifiable HCV RNA throughout the entire treatment period with at least 6 weeks of treatment, confirmed HCV RNA greater than the LLOQ after previously having unquantifiable HCV RNA, or a confirmed increase from nadir of at least one log10 in HCV RNA during treatment.
Time Frame: Up to 12 or 24 weeks after first dose
Population: Intent-to-treat population: all participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A | Arm B | Arm C
Number analyzed (Participants) | 100 | 31 | 29
percentage of participants | 1.0 [0.2 to 5.4] | 3.2 [0.6 to 16.2] | 3.4 [0.6 to 17.2]

4. Secondary Outcome: Percentage of Participants With Post-treatment Relapse Within 12 Weeks Following End of Treatment in Each Arm
Description: Post-treatment relapse was defined as defined as confirmed HCV RNA > LLOQ between the end of treatment and 12 weeks after the last dose of study drug among participants who completed treatment with HCV RNA < LLOQ at the end of treatment.
Time Frame: Up to 12 weeks after first dose
Population: Intent-to-treat population: all participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A | Arm B | Arm C
Number analyzed (Participants) | 98 | 30 | 28
percentage of participants | 3.1 [1.0 to 8.6] | 0.0 [0.0 to 11.4] | 0.0 [0.0 to 12.1]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) and serious adverse events (TESAEs) were collected from the time of study drug administration until 30 days after the last dose of study drug (up to 28 weeks).
Description: TEAEs and TESAEs are defined as any adverse event (AE) with an onset date that is after the first dose of study drug until 30 days after the last dose of study drug and were collected whether elicited or spontaneously reported by the participant.
Arm/Group | Arm A | Arm B | Arm C
Serious Adverse Events (participants affected / at risk) | 2/100 | 0/31 | 2/29
Other Adverse Events (participants affected / at risk) | 79/100 | 24/31 | 25/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (N=100) | Arm B (N=31) | Arm C (N=29)
OESOPHAGEAL VARICES HAEMORRHAGE (Gastrointestinal disorders) | 0 | 0 | 1
BILE DUCT STONE (Hepatobiliary disorders) | 0 | 0 | 1
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 0 | 0 | 1
APNOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (N=100) | Arm B (N=31) | Arm C (N=29)
ANAEMIA (Blood and lymphatic system disorders) | 8 | 2 | 4
NEUTROPENIA (Blood and lymphatic system disorders) | 5 | 0 | 1
PALPITATIONS (Cardiac disorders) | 4 | 0 | 2
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 19 | 2 | 3
CONSTIPATION (Gastrointestinal disorders) | 1 | 3 | 1
DIARRHOEA (Gastrointestinal disorders) | 5 | 3 | 2
DYSPEPSIA (Gastrointestinal disorders) | 17 | 4 | 5
NAUSEA (Gastrointestinal disorders) | 7 | 2 | 5
VOMITING (Gastrointestinal disorders) | 5 | 1 | 3
FATIGUE (General disorders) | 35 | 9 | 11
OEDEMA PERIPHERAL (General disorders) | 0 | 0 | 3
PYREXIA (General disorders) | 5 | 1 | 4
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 2 | 2 | 3
JAUNDICE (Hepatobiliary disorders) | 1 | 0 | 3
NASOPHARYNGITIS (Infections and infestations) | 13 | 0 | 2
SINUSITIS (Infections and infestations) | 2 | 0 | 2
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 0 | 2
BLOOD BILIRUBIN INCREASED (Investigations) | 0 | 1 | 2
HAEMOGLOBIN DECREASED (Investigations) | 5 | 2 | 2
DECREASED APPETITE (Metabolism and nutrition disorders) | 2 | 0 | 4
DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 | 0 | 2
HYPERURICAEMIA (Metabolism and nutrition disorders) | 8 | 4 | 2
BACK PAIN (Musculoskeletal and connective tissue disorders) | 5 | 2 | 0
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 2 | 2 | 2
DIZZINESS (Nervous system disorders) | 1 | 2 | 2
HEADACHE (Nervous system disorders) | 41 | 9 | 10
INSOMNIA (Psychiatric disorders) | 9 | 2 | 5
CHROMATURIA (Renal and urinary disorders) | 1 | 0 | 5
POLYURIA (Renal and urinary disorders) | 1 | 0 | 2
COUGH (Respiratory, thoracic and mediastinal disorders) | 6 | 4 | 9
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 1
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 3
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 3
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 1
PRURITUS (Skin and subcutaneous tissue disorders) | 23 | 4 | 9
RASH (Skin and subcutaneous tissue disorders) | 5 | 1 | 1
HYPERTENSION (Vascular disorders) | 1 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.